CLINICAL TRIAL: NCT05330793
Title: Randomized Double-blind, Placebo-controlled Trial on the Effects of an Oral Probiotic Intervention With or Without a Novel ADP-1 Toothpaste
Brief Title: The Effects of an Oral Probiotic Intervention With or Without a Novel ADP-1 Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Collaborators: Roseman University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202001
Record Dates: First submitted 2022-02-08; First posted 2022-04-15 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Oral Health
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled clinical study to evaluate the safety and efficacy of an oral probiotic intervention with or without a novel toothpaste and compared with placebo toothpaste and placebo lozenges.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- : Oral probiotic lozenges + placebo toothpaste (toothpaste without ADP-1) (Other): 1 active oral probiotic with placebo toothpaste
  Interventions: Dietary Supplement: Oral probiotic; Dietary Supplement: Placebo
- Oral probiotic lozenges + toothpaste with ADP-1 (Active Comparator): Oral probiotic and ADP1 toothpaste
  Interventions: Dietary Supplement: Oral probiotic
- Placebo lozenges (lozenges without oral probiotics) + placebo toothpaste (toothpaste without ADP-1) (Placebo Comparator): Placebo without oral probiotics or ADP1 toothpaste
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral probiotic — an oral probiotic intervention with or without a novel ADP1 toothpaste
  Other Names: ADP1 toothpaste
  Arms: : Oral probiotic lozenges + placebo toothpaste (toothpaste without ADP-1); Oral probiotic lozenges + toothpaste with ADP-1
Dietary Supplement: Placebo — placebo without Oral probiotic or toothpaste
  Arms: : Oral probiotic lozenges + placebo toothpaste (toothpaste without ADP-1); Placebo lozenges (lozenges without oral probiotics) + placebo toothpaste (toothpaste without ADP-1)

SUMMARY:
* Randomized double-blind, placebo-controlled trial on the effects of an oral probiotic intervention with or without a novel ADP-1 toothpaste Objective
* Determine the safety and effectiveness of oral probiotic intervention with or without a novel toothpaste and compare with placebo

DETAILED DESCRIPTION:
Hypotheses:

1. Subjects using oral probiotics will have better oral health than subjects using placebo toothpaste and placebo lozenges.
2. Subjects using oral probiotics and ADP-1 toothpaste will have better oral health than subjects using oral probiotics and regular toothpaste, and subjects using regular toothpaste and placebo lozenges.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65 years old
* Fluent in English
* Have mild to moderate gingivitis (i.e., probing depth between 3mm and 5mm)
* Bleeding on probing on 30%+ areas
* Able to perform oral hygiene adequately after formal instructions
* Able to understand and comply with study procedure
* Able to provide written informed consent
* Able to come to Roseman Dental Clinics in South Jordan for a 90-minute pre-screening to determine eligibility
* Able to complete five (90-minute) clinic visits in 2-week intervals

Exclusion Criteria:

* • Probing depths less than 3mm

  * Breastfeeding, pregnant or trying to become pregnant
  * Currently taking or have taken any of the following within 30 days of enrollment:

    * Oral probiotics
    * Antibiotic medications
    * Antifungal medications (e.g., nystatin, clotrimazole, ketoconazole, griseofulvin)
    * Antiseptic medications
    * Immunosuppressant and/or chemotherapeutic medications
    * Medications that could affect gum response measurement (e.g., calcium channel blockers, cyclosporin, anti-seizures like phenytoin and related drugs, anti-inflammatory agents)
  * Frequent alcohol consumption (> 2 drinks per day, or > 8 per week for women, or > 15 per week for men)
  * Use of marijuana (which can cause dry mouth or other conditions) or recreational drugs
  * Use of tobacco products including chewing tobacco and all types of cigarettes (e-cigarettes)
  * Known allergy to any product ingredient (ingredient list provided by USANA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Gingival Index | 8 weeks
  • Gingival Index measures gingival condition of the marginal and interproximal tissues (mesial, lingual, distal, facial) separately on the basis of 0 to 3 with 0=Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.
Plaque Index | 8 weeks
  • Plaque index is used as a method of recording the presence of plaque on individual tooth surfaces. These surfaces are mesial, distal, buccal and lingual.

SECONDARY OUTCOMES:
Halitosis | 8 weeks
  • Halitosis will be measured using a digital bad breath checker. The instrument is a small device with a sensor that sits near your mouth. This instrument senses volatile sulfur compounds or VSCs and produces a parts-per-billion (ppb) measurement of the foul-smelling compounds.
Intraoral Imaging | 8 weeks
  • Intraoral imaging of tooth decay can be measured in at least one of the following methods: (1) Using traditional intraoral imaging camera in the dental clinics to visualize tooth decay on the tooth surface, and (2) Using a laser fluorescence pen to detect tooth decay.
SAQ | 8 weeks
  Self-Assessment Questionnaire will consist of no more than 100 questions examining quality of life across one or several of these domains: (1) social well-being, (2) mental well-being, (3) physical well-being, (4) oral health and (5) dental hygiene and halitosis.dental hygiene and halitosis.
Microbial Community Analysis | 8 weeks
  Oral swabs from the gum line will be collected using DNA Genotek OMNIgene-ORAL swab kits and stored in the accompanying swab storage tube for microbial community analysis. qPCR testing will be performed in house in USANA.

CONTACTS AND LOCATIONS:
Locations (1):
- Roseman University of Health Sciences College of Dental Medicine, South Jordan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
YES